CLINICAL TRIAL: NCT06214286
Title: Adding Shock Wave Therapy to Kinesio Taping Improves Carpal Tunnel Syndrome in Physical Therapist Females. A Randomized Controlled Trial.
Brief Title: Adding Shock Wave Therapy to Kinesio Taping Improves Carpal Tunnel Syndrome in Physical Therapist Females.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Badr University (Other)
Responsible Party: Principal Investigator, Mina Magdy Wahba, Lecturer, Badr University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUCN1
Record Dates: First submitted 2023-12-11; First posted 2024-01-19 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Physiopathology
Keywords: Shockwave; Carpel tunnel

STUDY DESIGN:
Intervention Model Description: A total of 100 females patients ( two groups each group 50 females) who were diagnosed as having mild or moderate carpal tunnel syndrome were included in the study. One group received shock wave therapy with the conventional physical therapy program including kinesio taping, the second group received the conventional physical therapy program including kinesio taping without shock wave therapy. The patients were evaluated using a Visual Analog Scale-pain, a Visual Analog Scale-numbness, the Boston Symptom Severity Scale, the Boston Functional Status Scale, and handgrip strength tests and Nerve conduction study before treatment 1 and 12 wks after the treatment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shockwave (Experimental): One group received shock wave therapy with the conventional physical therapy program including kinesio taping
  Interventions: Device: Shockwave; Other: Kinesio taping; Other: conventional physical therapy
- conventional (Active Comparator): conventional physical therapy program including kinesio taping without shock wave therapy
  Interventions: Other: Kinesio taping; Other: conventional physical therapy

INTERVENTIONS:
Device: Shockwave — Shockwave therapy
  Arms: Shockwave
Other: Kinesio taping — Kinesio taping application
Other: conventional physical therapy — conventional physical therapy

SUMMARY:
PURPOSE: To investigate the effect of adding Shock wave therapy to kinesio taping on relieving carpal tunnel syndrome symptoms in physical therapist females.

BACKGROUND: shockwave therapy is a popular non-invasive therapeutic modality in the medical field for the treatment of numerous musculoskeletal disorders. Shockwaves can generate interstitial and extracellular responses, producing many beneficial effects such as: pain relief, vascularization, protein biosynthesis, cell proliferation, neuro and chondroprotection, and destruction of calcium deposits in musculoskeletal structures. shockwave combined with conventional physiotherapy is an effective noninvasive treatment for mild-to-moderate carpal tunnel syndrome that produces greater and longer-lasting results than conventional physiotherapy alone HYPOTHESES: Adding Shock wave therapy to kinesio taping has positive effects on carpal tunnel syndrome in physical therapist females.

RESEARCH QUESTION: Does adding Shock wave therapy to kinesio taping has positive effects on carpal tunnel syndrome in physical therapist females?

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 20 and 40 years
* diagnosed as having mild and moderate carpal tunnel syndrome through clinical parameters and nerve conduction studies (NCSs),

Exclusion Criteria:

- Having any systemic diseases such as renal failure, peptic ulcer, diabetes mellitus, hypothyroidism, coagulopathy, inflammatory rheumatic disease, having a cardiac pacemaker, cervical radiculopathy, polyneuropathy or brachial plexopathy, systemic corticosteroid use, fracture or trauma history in the forearm and wrist pregnancy and lactation, having received a carpal tunnel syndrome surgery, thoracic outlet syndrome or severe carpal tunnel syndrome.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | 1 and 12 week
  It is a self reported outcome which is a 10 cm line with zero at one end indicating no pain and 10 at the other end indicating maximum pain. Patient will be asked to mark the current pain on the scale and the distance from the starting point (0) will be measured

SECONDARY OUTCOMES:
Numbness Visual Analog Scale | 1 and 12 week
  It is self reported outcome, which is a 10 cm line with zero at one end indicating no numbness and 10 at the other end indicating maximum numbness.Patient will be asked to mark the current numbness on the scale, and the distance from the starting point (0) will be measured
Boston Carpal Tunnel Questionnaire | 1 and 12 week
  a Questionnaire widely used for assessing function and/or symptoms in patients with carpal tunnel syndrome. It consists of two separate scales: the Symptom Severity Scale (SSS), which consists of 11 questions and the Functional Status Scale (FSS), which consists of 8 items and requires respondents to score the difficulty of each item on a five-point scale. A final score is calculated for each scale (the sum of the individual scores divided by the number of items) and ranges from 1 to 5, with a higher score indicating a more severe handicap.
handgrip strength | 1 and 12 week
  hand grip strength will be measured by a hand held dynamometer Participants will be instructed to grip the dynamometer as strongly as they possibly can, using their affected hand. Three measurements will be taken and the highest value will be used in the analysis
electrodiagnostic study for median nerve | 1 and 12 week
  Sensory distal latency and motor distal latency of the median nerve will be measured by electromyography device according to standard protocol ( sensory distal latency stimulated at wrist and recorded 14cm at middle finger) and motor distal latency was stimulated at wrist and recorded from abductor pollicis brevis muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Omnya samy Abdallah Ghoneim, PhD, Study Chair — Department of Physical Therapy for Pediatrics and Pediatric Surgery, Faculty of Physical Therapy, Badr University in Cairo, Egypt.; Mina Magdy Wahba, PhD, Principal Investigator — Department of Physical Therapy for Orthpedics, Suez University; Fatma Said Zidan Hamed, PhD, Study Chair — Department of Physical therapy for Neuromuscular Disorders & its Surgery, Faculty of Physical Therapy, Badr University in Cairo, Egypt; Hanaa Samir Mohamed Abd el fatah, PhD, Study Director — Faculty of Physical therapy, Modern University for Technology and Information, Egypt.; Doha Hamed Moustafa Al-Afify, PhD, Study Chair — Basic Sciences Department, Faculty of Physical Therapy, Badr University in Cairo, Egypt; Doaa Saeed, Study Director — Department of Physical Therapy for Women's Health, Faculty of Physical Therapy, Badr University in Cairo, Cairo, Egypt
Locations (1):
- Badr University in Cairo (BUC), Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No